CLINICAL TRIAL: NCT01024959
Title: Clinical Evaluation of the PROGENSA(R) PCA3 Assay in Men With a Previous Negative Biopsy Result
Brief Title: Clinical Evaluation of the PROGENSA(Registered Trademark) Prostate Cancer Gene 3 (PCA3) Assay in Men With a Previous Negative Biopsy Result
Acronym: PCA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009PCA301
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Prostate Biopsy; PCA3
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCA3 Assay (Experimental)
  Interventions: Other: PCA3 Assay

INTERVENTIONS:
Other: PCA3 Assay — Post-Digital Rectal Exam (DRE) urine collected prior to prostate biopsy

SUMMARY:
The objective of this multi-center clinical study is to determine the association of the PCA3 Score with prostate biopsy outcome and validate the assay's performance characteristics in men with previous negative prostate biopsies. An elevated PCA3 Score is thought to be associated with an increased likelihood of positive biopsy. The results of this study are intended to be used for regulatory filings for use as an in vitro diagnostic test.

DETAILED DESCRIPTION:
PCA3 is a gene that is highly over-expressed in more than 90% of prostate cancers, and that can be quantified in urine specimens following a digital rectal examination. Studies have shown that because PCA3 is highly specific for prostate cancer, it predicts the results of repeat biopsies more accurately than traditional prostate-specific antigen (PSA) testing. Gen-Probe's PROGENSA(R) PCA3 assay is the first urine-based molecular diagnostic assay for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men 40+ years of age who have had at least 1 previous negative prostate biopsy, who have never had a positive prostate biopsy, and who have been recommended for a repeat biopsy by their clinician.
* The subject must be able to comprehend and sign an approved informed consent form and other applicable study enrollment documents

Exclusion Criteria:

* Use of medications or hormones that are known to affect serum PSA levels within 3 - 6 months of study enrollment
* Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment
* History of prostate cancer
* History of invasive treatments for benign prostatic hypertrophy (BPH) or lower urinary tract symptoms within 6 months of study enrollment
* Medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial, or constitutes an unacceptable risk to the subject
* Participation in pharmaceutical or treatment related clinical study within 6 months of study enrollment. Exception: Trials for non-prostate conditions may be acceptable, with approval by the investigator and Sponsor

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (13):
- United States (13):
  - HealthCare Partners Medical Group, Los Angeles, California
  - San Diego Clinical Trials, San Diego, California
  - South Florida Medical Research, Aventura, Florida
  - Specialists in Urology, Naples, Florida
  - Florida Urology Specialists, Sarasota, Florida
  - Metropolitan Urology, PSC, Jeffersonville, Indiana
  - Regional Urology Specialists, LLC, Shreveport, Louisiana
  - AccuMed Research Associates, Garden City, New York
  - TriState Urologic Services PSC Inc. dba The Urology Group, Cincinnati, Ohio
  - Columbus Urology Research, LLC, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia

REFERENCES:
- [Derived] Gittelman MC, Hertzman B, Bailen J, Williams T, Koziol I, Henderson RJ, Efros M, Bidair M, Ward JF. PCA3 molecular urine test as a predictor of repeat prostate biopsy outcome in men with previous negative biopsies: a prospective multicenter clinical study. J Urol. 2013 Jul;190(1):64-9. doi: 10.1016/j.juro.2013.02.018. Epub 2013 Feb 14. PMID 23416644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 507 male subjects were recruited from 14 clinical sites in the United States including academic institutions, community-based urology clinics and group health organizations.
Groups:
- Prostate Cancer Gene 3 (PCA3) Assay: PCA3 Assay : Post-Digital Rectal Exam (DRE) urine collected prior to prostate biopsy. N=495 represents the total number of subjects eligible for the study. 507 subjects were enrolled, 12 were determined to be ineligible.
Period: Overall Study
Arm/Group | Prostate Cancer Gene 3 (PCA3) Assay
Started | 507
Completed | 466
Not Completed | 41
Not completed — ineligible | 12
Not completed — results not evaluable | 12
Not completed — missing results required for analysis | 17

BASELINE CHARACTERISTICS:
Groups:
- PCA3 Assay: PCA3 Assay : Post-DRE urine collected prior to prostate biopsy. N=495 represents the total number of subjects eligible for the study. 507 subjects were enrolled, 12 were determined to be ineligible.
Arm/Group | PCA3 Assay
Number analyzed (Participants) | 495
Age Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 495
Region of Enrollment [Number; unit: participants]
  United States | 495

OUTCOME MEASURES:

1. Primary Outcome: Association of PCA3 Score With Prostate Biopsy Outcome (PCA3 Score Using Cutoff of 25.)
Description: The likelihood of positive biopsy was determined by the PCA3 Score expressed as a binary categorical variable: PCA3 Score >=25 was positive, PCA3 Score <25 was negative
Time Frame: At the time of biopsy
Population: A total of n=466 subjects have valid and reportable PCA3 Scores and disease status (determined by biopsy result), and who were 50 years of age or older.
Measure: Number; unit: participants
Groups:
- PCA3 Assay: PCA3 Assay : Post-DRE urine collected prior to prostate biopsy
- Subjects With Positive Biopsy Result: Presence of prostate cancer defined by one or more positive biopsy cores
- Subjects With Negative Biopsy Result: Absence of prostate cancer defined by no positive biopsy cores (note: presence of high grade PIN and/or atypia are classified as negative biopsy results)
Arm/Group | PCA3 Assay | Subjects With Positive Biopsy Result | Subjects With Negative Biopsy Result
Number analyzed (Participants) | 466 | 102 | 364
participants
  All PCA3 Scores | 466 | 102 | 364
  PCA3 Score >=25 | 235 | 79 | 156
  PCA3 Score <25 | 231 | 23 | 208

ADVERSE EVENTS:
Description: Our definition of at risk population is any unique subject who gave a post-digital rectal exam (DRE) urine sample, regardless of eligibility(n=498 of n=507 participants who started the study). n=106 of these subjects had a positive biopsy; n=389 had negative biopsy; n=3 had no biopsy.
Arm/Group | PCA3 Assay | Subjects With Positive Biopsy Result | Subjects With Negative Biopsy Result | Subjects With no Biopsy Performed
Serious Adverse Events (participants affected / at risk) | 0/498 | 0/106 | 0/389 | 0/3
Other Adverse Events (participants affected / at risk) | 0/498 | 0/106 | 0/389 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less